CLINICAL TRIAL: NCT05052359
Title: Aberrant Helix Pomatia Agglutinin Binding Glycan Expression Changes With the Phenotype of Follicular Thyroid Tumours
Brief Title: Aberrant Helix Pomatia Agglutinin Binding Glycan Expression in Follicular Thyroid Tumours
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Rajeev Parameswaran, Asst. Prof. Rajeev Parameswaran FRCSI MPhil FRCS FAMS, National University Health System, Singapore
Other Study IDs: 2014/00378
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Follicular Thyroid Cancer
Keywords: Glycosylation
MeSH Terms: conditions — Adenocarcinoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lectin-histochemistry retrospectively performed — Lectin-histochemistry was performed on 37 archival paraffin wax-embedded specimens of various follicular thyroid tumours (10 follicular adenomas (FA), 10 minimally invasive follicular carcinomas (miFTC), 13 widely invasive follicular cancers (wiFTC) and 4 metastatic follicular thyroid cancers (metFTC)).

SUMMARY:
Aberration of glycosylation is a hallmark of cancer cells, and plays an important role in oncogenesis and cancer progression, including metastasis. One of the markers of aberrant glycosylation (O-linked) is the binding of the lectin Helix pomatia agglutinin (HPA), which has been demonstrated in a wide range of human cancers, especially in tumours with a more aggressive phenotype. Data on the role of HPA within follicular neoplasms of the thyroid gland are currently lacking, therefore we sought to investigate possible changes in cell surface glycosylation associated with this type of neoplasms.

DETAILED DESCRIPTION:
Lectin-histochemistry was performed on 37 archival paraffin wax-embedded specimens of various follicular thyroid tumours (10 follicular adenomas (FA), 10 minimally invasive follicular carcinomas (miFTC), 13 widely invasive follicular cancers (wiFTC) and 4 metastatic follicular thyroid cancers (metFTC)). Sections were scored as positive when ≥5% of cancer cells labelled positive, and scored as negative when <5% labelled positive for HPA binding. Assessments of HPA-binding were performed by two observers, who were blinded to the identity of the sample, and their results were compared.

ELIGIBILITY:
Inclusion Criteria:

* For this retrospective cohort study, 37 patients who underwent thyroid surgery for a thyroid follicular neoplasm between 2005 and 2018 were identified from our institutional database and their tumours, characteristics and outcomes were analysed.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For this retrospective cohort study, 37 patients who underwent thyroid surgery for a thyroid follicular neoplasm between 2005 and 2018 were identified from our institutional database and their tumours, characteristics and outcomes were analysed.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Positivity of HPA-labelling | between 2005 and 2018
  Difference in HPA-binding among the phenotype of follicular lesions - percentage of positively labelled cancer cells: positive = ≥5% of cancer cells labelled positive

SECONDARY OUTCOMES:
HPA-binding and other tumor markers | between 2005 and 2018
  A Statistical association of HPA-binding positivity with other known adverse prognostic tumour markers (e.g. capsular or lymphovascular invasion) will be assessed using crosstabs and the non-parametric product limit method. Binary logistic regression models will be further developed using relevant clinicopathologic variables to determine their association with HPA-labelling to produce relative risks (odds ratios (ORs)).

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No